CLINICAL TRIAL: NCT03850691
Title: A Phase 2 Study of Palliative Radiation and Combination Sequential Immunotherapy for Metastatic Cutaneous Melanoma and Ocular Melanoma
Brief Title: Radiation and Combination Immunotherapy for Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018LS110
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Melanoma
Keywords: MM
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; Administration, Cutaneous; Vision, Ocular

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Nivolumab (Experimental)
  Interventions: Drug: Aldesleukin: All Patients; Drug: Nivolumab: Cohort 1 (Cutaneous)
- Cohort 2: Nivolumab & Ipilimumab (Experimental)
  Interventions: Drug: Aldesleukin: All Patients; Drug: Nivolumab: Cohort 2 (Ocular); Drug: Ipilimumab: Cohort 2 (Ocular)

INTERVENTIONS:
Drug: Aldesleukin: All Patients — Cycle 1:
  (600,000 U/kg/dose) given as a bolus infusion once every 8 to 12 hours over 5 days or until no longer tolerated (to a maximum of 10 doses). Administered as an inpatient.
  Days 1-5 and Days 15-19 (all patients)
  Other Names: IL-2
Drug: Nivolumab: Cohort 1 (Cutaneous) — Cycle 1: 6 Week Duration Nivolumab 240 mg IV
  Cycle 2: 6 Week Duration Nivolumab 240 mg IV on Day 1, 15 and 29
  Cycle 3: 4 Week Duration Nivolumab 240 mg IV on Day 1 and 15
  Patients may continue maintenance nivolumab 240 mg IV every 2 weeks OR nivolumab 480 mg IV every 4 weeks per 2018 FDA approval at discretion of the treating physician and independent of this study
  Arms: Cohort 1: Nivolumab
Drug: Nivolumab: Cohort 2 (Ocular) — Cycle 1: 6 Week Duration Nivolumab 3 mg/kg IV on Day 29
  OR for a high risk patient with an excellent performance status, the following regimen may be given at the discretion of the treating investigator:
  Nivolumab 1 mg/kg IV on Day 29
  Cycle 2: 6 Week Duration Nivolumab on Day 8 and on Day 29 using the same dose regimen as used Cycle 1 Day 29
  Cycle 3: 4 Week Duration Nivolumab on Day 8 using the same dose regimen as used Cycle 1 Day 29.
  Patients may continue maintenance nivolumab 240 mg IV every 2 weeks OR nivolumab 480 mg IV every 4 weeks per 2018 FDA approval at discretion of the treating physician and independent of this study
  Arms: Cohort 2: Nivolumab & Ipilimumab
Drug: Ipilimumab: Cohort 2 (Ocular) — Cycle 1: 6 Week Duration Ipilimumab 1 mg/kg IV on Day 29
  OR for a high risk patient with an excellent performance status, the following regimen may be given at the discretion of the treating investigator:
  Ipilimumab 3 mg/kg IV on Day 29
  Cycle 2: 6 Week Duration Ipilimumab on Day 8 and on Day 29 using the same dose regimen as used Cycle 1 Day 29
  Cycle 3: 4 Week Duration Ipilimumab on Day 8 using the same dose regimen as used Cycle 1 Day 29
  Arms: Cohort 2: Nivolumab & Ipilimumab

SUMMARY:
This is a Phase 2 study designed to evaluate the combination of checkpoint blockade and aldesleukin (IL-2) therapy after a course of standard of care palliative radiation in the management of unresectable metastatic melanoma. To be eligible, a patient must have a minimum of 3 (preferably >5) radiographically distinct, measurable (>1.5 cm) lesions based on RECIST 1.1. Metastatic cutaneous melanoma must be refractory to standard immunotherapy drugs, molecular targeted agents and/or chemotherapy. Patients with ocular melanoma subtypes may enroll in this study without prior therapy, as there is no standard front-line therapy for this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven unresectable, metastatic melanoma refractory to standard immunotherapy drugs or regimens, including prior treatment with Aldesleukin (IL-2), GM-CSF, Ipilimumab, Nivolumab, Pembrolizumab, and/or Imlygic (T- VEC).

  * Prior clinical trial participation or treatment with molecularly targeted agents (i.e. Vemurafenib/Cobimetinib, Dabrafenib/Trametinib) or chemotherapy (i.e. Temozolomide, Dacarbazine, Platinum, or Taxanes) is permitted.
  * Patients with ocular melanoma may enroll (Cohort 2) without prior therapy as there is no standard 1st line therapy for this subset of melanoma.
* Must have a minimum of 3 radiographically distinct (>1.5 cm) lesions measurable by RECIST 1.1 at time of study enrollment (>5 preferred).

  * A maximum of 2 metastases per treated organ may be targeted for palliative radiation, but must be separated by more than 5 cm of normal tissue
  * At least 2 non-irradiated lesions are required for systemic response assessments
* Pulmonary metastases: Pulmonary metastasis permissible. Appropriate candidates with lung lesions may be considered for ablative hypofractionation using SBRT.
* Hepatic metastases: Hepatic metastasis permissible. Appropriate candidates with metastasis to liver may be considered for ablative hypofractionation using SBRT .
* Brain metastases: Brain metastases may be treated using Gamma Knife Radiosurgery (GKR) or whole brain radiation therapy (WBRT) per the treating radiation oncologist. Total radiation dose and number of fractions will be determined by the treating radiation oncologist based on anatomic and dosing constraints. MRI of the vertebral column is required for all patients with suspected epidural tumor extension.
* Must have sufficient archival tissue block material (1.5 x 1.5 x 1.5 cm) and/or newly obtained core or excisional biopsy of tumor tissue; minimum of 2 cores.
* ECOG performance status 0 or 1 (Appendix 2)
* Age 18 through 80 years of age; > 80 years of age must be approved by Principal Investigator.
* Adequate organ function within 14 days of enrollment (30 days for pulmonary and cardiac assessments) defined as:

  * Hematologic: leukocytes ≥ 2,000/mcL, ANC ≥ 1,000/mcL, hemoglobin ≥ 9.0 g/dL, platelets ≥ 100,000/mcL unsupported by transfusions
  * Renal: Serum creatinine ≤ 1.8 mg/dL; for patients with a creatinine > 1.5 mg/dL or a history of renal dysfunction, an estimated glomerular filtration rate ≥ 35 mL/min/1.73 m2 is required
  * Hepatic: AST, ALT, and alkaline phosphatase ≤ 5 x upper limit of normal and total bilirubin ≤ 2.0 mg/dL
  * Pulmonary: oxygen saturation ≥90% on room air; corrected DLCO and FEV1, ≥ 60% predicted
  * Cardiac: Absence of clinical decompensated congestive heart failure or uncontrolled arrhythmia; left ventricular ejection fraction (echocardiogram within 6 months permitted) ≥ 40%. QTc must be < 450 ms in males and < 470 ms in females.
* A minimum of 1 week between last anti-tumor treatment if given, and 1st dose of radiation therapy (not applicable for patients enrolling after palliative radiation therapy).
* Recovery from previous cancer treatment if applicable defined as ≤ Grade 1 (by CTCAE 5.0 criteria) at enrollment
* Women of childbearing potential and males with partners of childbearing potential must agree to the use of barrier methods of contraception, hormonal contraceptives, or abstain from heterosexual activity for the duration of study treatment and for 3 months after the last dose of study drug.
* Ability to understand and provide voluntary written consent

Exclusion Criteria:

* Pregnant or breast feeding. The agents used in this study have the potential to harm a fetus. Radiation is a known teratogen. There is insufficient information regarding potential for fetal harm during immunotherapy at this time. Biological females of childbearing potential must have a negative pregnancy test within 14 days of enrollment.
* Concurrent use of high dose steroids; chronic steroid use of < 2 mg dexamethasone or equivalent per day is permissible
* Concurrent malignancy requiring active treatment, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ
* Severe and active autoimmune diseases requiring systemic immunosuppression
* Prior organ allograft or allogeneic transplantation
* Other contraindication to IL-2, nivolumab, ipilimumab, or combination immunotherapy per treating medical oncologist
* Live vaccines within 30 days prior to the first dose of IL-2 and while participating in the trial. Examples of live vaccines include, but are not limited to, measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally inactivated virus vaccines and are allowed. Intranasal influenza vaccine (eg, Flu - Mist®) is a live attenuated vaccine, and is not allowed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evidio Domingo-Musibay, MD, Principal Investigator — Division of Hematology, Oncology and Transplantation, University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Burnsville, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Nivolumab: Aldesleukin: All Patients: Cycle 1:
  (600,000 U/kg/dose) given as a bolus infusion once every 8 to 12 hours over 5 days or until no longer tolerated (to a maximum of 10 doses). Administered as an inpatient.
  Days 1-5 and Days 15-19 (all patients)
  Nivolumab: Cohort 1 (Cutaneous): Cycle 1: 6 Week Duration Nivolumab 240 mg IV
  Cycle 2: 6 Week Duration Nivolumab 240 mg IV on Day 1, 15 and 29
  Cycle 3: 4 Week Duration Nivolumab 240 mg IV on Day 1 and 15
  Patients may continue maintenance nivolumab 240 mg IV every 2 weeks OR nivolumab 480 mg IV every 4 weeks per 2018 FDA approval at discretion of the treating physician and independent of this study
- Cohort 2: Nivolumab & Ipilimumab: Aldesleukin: All Patients: Cycle 1:
  (600,000 U/kg/dose) given as a bolus infusion once every 8 to 12 hours over 5 days or until no longer tolerated (to a maximum of 10 doses). Administered as an inpatient.
  Days 1-5 and Days 15-19 (all patients)
  Nivolumab: Cohort 2 (Ocular): Cycle 1: 6 Week Duration Nivolumab 3 mg/kg IV on Day 29
  OR for a high risk patient with an excellent performance status, the following regimen may be given at the discretion of the treating investigator:
  Nivolumab 1 mg/kg IV on Day 29
  Cycle 2: 6 Week Duration Nivolumab on Day 8 and on Day 29 using the same dose regimen as used Cycle 1 Day 29
  Cycle 3: 4 Week Duration Nivolumab on Day 8 using the same dose regimen as used Cycle 1 Day 29.
  Patients may continue maintenance nivolumab 240 mg IV every 2 weeks OR nivolumab 480 mg IV every 4 weeks per 2018 FDA approval at discretion of the treating physician and independent of this study
  Ipilimumab: Cohort 2 (Ocular): Cycle 1: 6 Week Duration Ipilimumab 1 mg/kg IV on Day 29
  OR for a high risk patient with an excellent performance status, the following regimen may be given at the discretion of the treating investigator:
  Ipilimumab 3 mg/kg IV on Day 29
  Cycle 2: 6 Week Duration Ipilimumab on Day 8 and on Day 29 using the same dose regimen as used Cycle 1 Day 29
  Cycle 3: 4 Week Duration Ipilimumab on Day 8 using the same dose regimen as used Cycle 1 Day 29
Period: Overall Study
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab & Ipilimumab
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab & Ipilimumab | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Determine the objective response rate (ORR). The ORR will be presented as the proportion of patients who achieved complete response (CR) or partial response (PR). In general, categorical data measurements will be summarized as counts and percentages (or proportions). The disease control rate (DCR) will be presented as the proportion of patients with CR, PR, or stable disease. The best overall response (BOR) will be measured as the maximum change from baseline in the sum of the longest diameter for each of the target lesions over the full 2 year follow-up period.
Time Frame: up to approximately 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab & Ipilimumab
Number analyzed (Participants) | 1 | 3
Participants | 1 | 1

2. Primary Outcome: Safety and Tolerability of Sequential Combination Immunotherapy (Incidence of Adverse Events)
Description: This will be achieved by the number of adverse event (AE) reports. AEs, SAEs, deaths, and abnormal laboratory values will be summarized by the proportion of patients who experience them. Descriptive statistics of safety will be presented using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All on-study AEs, Grade 3-4 AEs, treatment-related AEs, Grade 3-4 treatment-related AEs, SAEs, treatment-related SAEs, and AEs leading to discontinuation will be tabulated using the worst grade per NCI CTCAE v 5.0 criteria by system organ class.
Time Frame: Approximately up to 2 Years
Measure: Number; unit: Adverse events
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab & Ipilimumab
Number analyzed (Participants) | 1 | 3
Adverse events | 3 | 0

3. Primary Outcome: Safety and Tolerability of Sequential Combination Immunotherapy (Incidence of Stopping Rule Events)
Description: This will be measured by the number of participants who are suspended from the trial as noted by a stopping rule event. These events are determined after serious adverse events are graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The following events count toward an early stopping rule event: 1) Any Grade 2 or greater drug-related uveitis, eye pain, or blurred vision that does not respond to topical therapy and does not improve to Grade 1 severity within 7 days of checkpoint inhibitor OR requires systemic treatment with corticosteroids, 2) Any Grade 3 or greater non-skin, drug-related adverse event lasting > 7 days, including uveitis, pneumonitis, bronchospasm, diarrhea, colitis, neurologic toxicity, hypersensitivity reactions, and infusion reactions. In addition, the trial would be stopped and re-evaluated if there is ≥ 1 treatment-related mortality event.
Time Frame: Approximately up to 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab & Ipilimumab
Number analyzed (Participants) | 1 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From first visit dose to end of trial visit (16 weeks if received all cycles). The end of trial visit date is approximately 4 weeks after the last dose of the study drug. Follow-up for disease status and survival will continue for up to 2 years from study enrollment by electronic/phone contact every 3 months (± 2 weeks) unless the patient withdraws consent. This gives an approximate timeline of up to 2 years, as the survival status at 2 years could potentially include death as an SAE.
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab & Ipilimumab
All-Cause Mortality (participants affected / at risk) | 1/1 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Nivolumab (N=1) | Cohort 2: Nivolumab & Ipilimumab (N=3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — failure to thrive.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Nivolumab (N=1) | Cohort 2: Nivolumab & Ipilimumab (N=3)
Lymphocyte count decreased (Investigations) | 1 (1) | 0
Infections and infestations - Other, specify (Investigations) | 1 (1) | 0
Investigations - Other, specify (Investigations) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT03850691/Prot_SAP_000.pdf